CLINICAL TRIAL: NCT04606537
Title: Phase 1, Open-label, Parallel, 2-arm, Fixed-sequence Study to Investigate the Effect of Coadministration of CYP3A4 Inhibitor and CYP3A4 Inducer on the Pharmacokinetics, Safety, and Tolerability of KBP-5074 in Healthy Subjects
Brief Title: Drug to Drug Interaction Study of KBP-5074 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KBP5074-1-008
Record Dates: First submitted 2020-10-16; First posted 2020-10-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Drug Drug Interaction
Keywords: KBP5074; Healthy Subjects; itraconazole; rifampin
MeSH Terms: interventions — Itraconazole; Rifampin; KBP-5074

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Effects of CYP3A4 inhibition on KBP-5074) (Experimental)
  Interventions: Drug: Itraconazole; Drug: KBP-5074
- Cohort 2 (Effects of CYP3A4 induction on KBP-5074) (Experimental)
  Interventions: Drug: Rifampin; Drug: KBP-5074

INTERVENTIONS:
Drug: Itraconazole — 200 mg itraconazole, given orally as 20 mL × 10-mg/mL solution BID on Day 15, followed by QD dosing on Days 16 through 23, inclusive.
  Arms: Cohort 1 (Effects of CYP3A4 inhibition on KBP-5074)
Drug: Rifampin — 600 mg rifampin, given orally as 2 × 300-mg capsules QD on Days 15 through 25, inclusive.
  Arms: Cohort 2 (Effects of CYP3A4 induction on KBP-5074)
Drug: KBP-5074 — 0.5 mg KBP-5074, given orally as 1 × 0.5-mg tablet on Days 1 and 19 or Days 1 and 21

SUMMARY:
Open-label, parallel, 2-arm, fixed-sequence study to investigate the effect of coadministration of a CYP3A4 inhibitor (Cohort 1, itraconazole multiple dose) and CYP3A4 inducer (Cohort 2, rifampin multiple dose) on the plasma PK of a single dose of KBP-5074 in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 60 years of age, inclusive, at screening.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations

Exclusion Criteria:

* Significant history or clinical manifestation of any medical history, as determined by the investigator not appropriate to participate in this study.
* Use of any drugs or substances known to be strong or moderate inhibitors or inducers of CYP3A4 within 30 days prior to study drug administration. Medications will be reviewed by the medical monitor to determine acceptability for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter: Maximum observed concentration (Cmax) | Days 1 and 19 at predose (Cohort 1) and Days 1 and 21 at predose (Cohort 2) and at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 240 hours postdose.
  Maximum observed concentration (Cmax) - Plasma
Pharmacokinetic Parameter: Area under the concentration-time curve from time 0 to infinity (AUC0-∞) | Days 1 and 19 at predose (Cohort 1) and Days 1 and 21 at predose (Cohort 2) and at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 240 hours postdose.
  Area under the concentration-time curve from time 0 to infinity (AUC0-∞) - Plasma
Pharmacokinetic Parameter: Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) | Days 1 and 19 at predose (Cohort 1) and Days 1 and 21 at predose (Cohort 2) and at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168, and 240 hours postdose.
  Area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC0-tlast) - Plasma

CONTACTS AND LOCATIONS:
Overall Officials: James McCabe, Study Director — KBP Biosciences
Locations (1):
- QPS Missouri, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No